CLINICAL TRIAL: NCT00696345
Title: Feasibility Study for Performance of Septin 9 in Plasma From Cases With Colorectal Cancer and Controls With Non-Diseased, Non-Colorectal Disease and Non-Colorectal Cancers
Brief Title: Detection of Colorectal Cancer in Peripheral Blood by Septin 9 DNA Methylation Assay
Status: Completed | Type: Observational
Sponsor: Epigenomics, Inc (Industry)
Responsible Party: Michael Wandell VP Clinical, Regulatory, Quality, Epigenomics
Other Study IDs: Septin-9-2006
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; screening; biomarker; plasma; blood
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual plasma samples retained according to protocol.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Colorectal cancer patients, Stages I-IV
- 2: Non colorectal cancer patients, verified by colonoscopy

SUMMARY:
Epigenomics is developing a colon cancer screening assay based on differential methylation of specific CpG sites for the detection of early stage disease. A genome-wide methylation analysis and oligonucleotide array study using DNA from various stages of colon cancer and normal tissue have been completed to obtain candidate CpG markers. Based on results obtained in the above studies, Epigenomics has moved to the final stages of feasibility with a specific, highly sensitive real-time marker assay that is able to detect colon cancer DNA in blood plasma.

DETAILED DESCRIPTION:
From public health as well as health economics perspectives, the poor adoption of current screening options limits the effectiveness of CRC screening initiatives; as stated by Sidney Winawer, MD, "the best test is the one that gets done." Current CRC screening guidelines include FOBT, sigmoidoscopy (alone or with FOBT), or colonoscopy. Non-invasive screening is conducted using FOBT, which while inexpensive, exhibits a low compliance rate (around 16% in the US) due to its use restrictions, perceived inconvenience and lack of consumer acceptance. The gold standard procedure for CRC detection is colonoscopy; it exhibits excellent performance characteristics, but has a limited utility as a first line screen due to its high cost, healthcare delivery resource limitations, and inadequate patient acceptance. It is believed a noninvasive, first-line screening assay capable of detecting individuals with colorectal disease, confirmed by colonoscopy, would have greater utility for population screening.

Epigenomics has identified methylated gene regions that are specific for colorectal cancer or pre-malignant tissue. Aberrantly methylated genes represent attractive candidate markers for cancer screening, as cancer-specific methylation changes occur early in tumorigenesis, appear to be stable, yield a positive amplifiable signal, and can be assayed with high analytical sensitivity. Since methylation occurs early and in distinct genomic areas, it is possible to achieve high clinical sensitivity with a small number of methylated DNA markers. Studies have shown that aberrantly methylated DNA markers can be detected in tissue and body fluids and are highly correlated to colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 diagnosis of colorectal cancer

Exclusion Criteria:

* Group 2 diagnosis of colorectal cancer

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are identified at colonoscopy as having or not having colorectal cancer. Blood from all subjects was drawn either before or more than 2 days and up to 6 months after colonoscopy and prior to starting any cancer specific treatment. Cancer diagnosis was confirmed histologically from the surgical specimen and only adenocarcinomas were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2005-01; Primary Completion 2006-10 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Lofton-Day, PhD, Principal Investigator — Epigenomics, Inc
Locations (5):
- Germany (4):
  - Department of Surgery and Surgical Oncology, Charité Campus Berlin Buch, Berlin
  - Department of Visceral-, Thoracic- and Vascular Surgery, University Hospital Carl Gustav Carus, Dresden
  - Department of Surgery, University Hospital Schleswig-Holstein, Campus Lübeck, Lübeck
  - Völklingen Clinic, Völklingen
- Semmelweis University, Budapest, Hungary